CLINICAL TRIAL: NCT04948307
Title: A Randomized, Open-label, Parallel-group Study to Evaluate the Efficacy of the Digital Therapeutic OXD01 (MODIA™) in Combination With Sublingual Buprenorphine/Naloxone for the Treatment of Opioid Use Disorder
Brief Title: OXD01 in Combination With Sublingual Buprenorphine/Naloxone for Treatment of Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orexo AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXD01-001
Record Dates: First submitted 2021-06-22; First posted 2021-07-01 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Opioid-use Disorder
Keywords: digital therapy; cognitive behavioral therapy (CBT)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sublingual buprenorphine/naloxone (SL BUP/NAL) standard of care (SOC) background therapy (Other): Standard of care. Subjects in both groups will receive the assigned treatment for 24 weeks. Subjects in both groups may also be encouraged to participate in behavioral health therapies in accordance with the Investigator's standard of practice.
  Interventions: Other: Standard of Care
- Sublingual buprenorphine/naloxone (SL BUP/NAL) + OXD01 (Experimental): Standard of care + OXD01 (digital therapy). Subjects in both groups will receive the assigned treatment for 24 weeks. Subjects in both groups may also be encouraged to participate in behavioral health therapies in accordance with the Investigator's standard of practice.
  Interventions: Device: OXD01 digital therapy; Other: Standard of Care

INTERVENTIONS:
Device: OXD01 digital therapy — OXD01 digital therapy, 1-2 times per week 15-30 minutes each time.
  Arms: Sublingual buprenorphine/naloxone (SL BUP/NAL) + OXD01
Other: Standard of Care — Sublingual buprenorphine/naloxone Medication-assisted treatment, the current standard for opioid addiction; the use of medications in combination with counseling

SUMMARY:
This is an open-label, randomized, parallel-group multicenter study designed to evaluate the efficacy of the digital therapeutic OXD01 (MODIA) combined with sublingual buprenorphine/naloxone standard of care (SL BUP/NAL SOC) background therapy compared to SL BUP/NAL alone to change opioid use patterns in subjects with opioid use disorder (OUD).

Approximately 400 subjects will be randomized. The study will include a screening visit and a randomization visit, followed by 24 weeks of study treatment. Subjects will be scheduled for evaluation visits, which will include a urine drug screen (UDS) and a self-report of drug use, weekly during the first four weeks of treatment, then every other week from weeks 5 through 12, then monthly through week 25. Subjects will also return to the site for only a UDS and a self-report of drug use each week between the evaluation visits.

The primary objective of the study is to determine whether the combination of sublingual (SL) buprenorphine/naloxone (BUP/NAL) standard of care (SOC) background therapy and the digital therapeutic OXD01 is superior to SL BUP/NAL alone to reduce opioid use.

DETAILED DESCRIPTION:
Medication-assisted treatment, the current standard for opioid addiction, is the use of medications in combination with counseling and behavioral therapies to provide a "whole-patient" approach to the treatment of OUD. However, patients may not have optimal access to face-to-face clinical behavioral health services. Digital therapeutics can help bridge the gap between accessible services and optimal treatment of OUD, the primary goal of which is to reduce the use of opioids. OXD01 is a device-based digital therapeutic, designed to offer individuals diagnosed with OUD quality psychotherapy intervention based on cognitive behavioral therapy and motivational interviewing. This study is being conducted to determine the value of OXD01 when combined with medication to change opioid use patterns in subjects with OUD.

Note: No investigational product will be administered as part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 - 65 years of age at the screening visit, fluent in English and able to read, comprehend, and willingly sign the informed consent form (ICF).
2. Voluntarily seeking treatment for OUD.
3. In the judgment of the Investigator has the appropriate hearing, vision, manual dexterity, ability to understand instructions, and ability to use and understand internet-based applications.
4. Currently meets the criteria for moderate or severe opioid use disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-V (Appendix B).
5. Has a positive UDS for opioids at screening that is consistent with their drug use history.
6. In good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
7. Agrees not to take any buprenorphine products other than those prescribed by the Investigator during participation in the study, and agrees to use OXD01 as directed if randomized to that treatment group.
8. Completed SL BUP/NAL induction, with physical withdrawal symptoms reduced so the subject is able to fulling participate in OXD01 training, if randomized to that treatment group, and is no greater than 14 days from the first dose of SL BUP/NAL induction.

Exclusion Criteria:

* 1. Unwilling or unable to comply with the requirements of the protocol or are in a situation or condition that, in the opinion of an Investigator, may interfere with participation in the study (e.g., does not have reliable internet access).

  2. History of allergy or sensitivity to naloxone, buprenorphine or other opioids, or history of any drug hypersensitivity or intolerance which, in the opinion of an Investigator, would compromise the safety of the subject.

  3. Used an investigational drug within 30 days or 5 half-lives (whichever is greater) prior to randomization.

  4. Received prescribed medication-assisted treatment with buprenorphine, methadone, or naltrexone for opioid use disorder within 14 days prior to screening.

  5. Past or present diseases that, judged by an Investigator and based on available medical history/records, may jeopardize the safety of the subject or impact the validity of the study results.

  6. Tongue piercing, or piercings in the mouth or oral deformities that may affect sublingual absorption, in the opinion of an Investigator.

  7. Hospitalization for a psychiatric disorder in the past 30 days, not including inpatient treatment for drug rehabilitation.

  8. Schizophrenia, or other serious mental illness defined as a mental, behavioral, or emotional disorder resulting in serious functional impairment which substantially interferes with or limits participation in the study.

  9. A Quick Inventory of Depression Symptoms - Self-Report (QIDS-SR, Appendix C) score ≥ 16 (severe depression) or a rating of 2 or 3 for question 12 (Thoughts of Death or Suicide) at screening.

  10. A current diagnosis, other than opioid use disorder, requiring chronic opioid treatment.

  11. Chronic pain that is unremitting or unstable. 12. Current DSM-V diagnosis of moderate to severe substance use disorder for psychoactive substances other than opioids, caffeine, marijuana, or nicotine.

  13. Requires current use of medications that are strong inhibitors or inducers of cytochrome P450 (CYP) 3A4 (Section 4.3.1).

  14. Any pending legal action that could affect participation or compliance in the trial.

  15. Is an employee of the Investigator or the trial site, with direct involvement in the proposed trial or other trials under the direction of the Investigator or trial site, or is a family member of the Investigator or an employee.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Capano, PharmD, Study Director — Orexo US, Inc.
Locations (21):
- United States (21):
  - Parkway Medical Center, Birmingham, Alabama
  - North County Clinical Research, Oceanside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Wetlin Research Associates, Inc, San Diego, California
  - Humanity Clinical Research, Pembroke Pines, Florida
  - Southern Illinois Associates LLC, Glen Carbon, Illinois
  - Otrimed Clinical Research, Edgewood, Kentucky
  - Patient First Medical Clinic, Dearborn, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - PsychCare Consultants Research, St Louis, Missouri
  - Dr. Vando Medical Services PC, The Bronx, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Neuro-Behavioral Clinical Research Center, North Canton, Ohio
  - CincyScience, West Chester, Ohio
  - Pahl Pharmaceuticals Professions, Oklahoma City, Oklahoma
  - Thalia Medical Center, Haverford, Pennsylvania
  - MD Medical Management, Kingston, Pennsylvania
  - Medically Assisted Recovery Service, Philadelphia, Pennsylvania
  - Institute of Addiction Medicine, Plymouth Meeting, Pennsylvania
  - Aspen Clinical Research, Orem, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 30 June 2021 to 12 April 2023 at 36 outpatient sites in the United States.
Pre-assignment Details: Screening All Consented Subjects
  n (%)
  Screened: 672 Screen failure: 235 ( 35.0) Primary reason for screen failure due to COVID-19: 2 ( 0.3)
  Primary reason for screen failure:
  Failure to meet randomization criteria - 134 ( 19.9) Lost to follow-up - 63 ( 9.4) Withdrawal by subject - 23 ( 3.4) Adverse event - 2 (0.3) Physician decision - 1 (0.1) Other - 11 (1.6) Missing - 1 (0.1)
Groups:
- SL BUP/NAL SOC Background Therapy: Sublingual buprenorphine/naloxone titrated to a maintenance dose that suppresses withdrawal signs and symptoms
  Subjects in both groups will receive the assigned treatment for 24 weeks. Subjects in both groups may also be encouraged to participate in behavioral health therapies in accordance with the Investigator's standard of practice.
- SL BUP/NAL SOC Background Therapy + OXD01: Sublingual buprenorphine/naloxone titrated to a maintenance dose that suppresses withdrawal signs and symptoms plus OXD01 digital therapy, accessed for 15-30 minutes, 1-2 times per week
  Subjects in both groups will receive the assigned treatment for 24 weeks. Subjects in both groups may also be encouraged to participate in behavioral health therapies in accordance with the Investigator's standard of practice.
Period: Overall Study
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Started | 218 | 219
Completed | 120 | 114
Not Completed | 98 | 105

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01 | Total
Number analyzed (Participants) | 218 | 219 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.41) | 41.9 (10.63) | 40.9 (010.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 111 | 201
  Male | 128 | 108 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 41 | 78
  Not Hispanic or Latino | 171 | 167 | 338
  Unknown or Not Reported | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 30 | 25 | 55
  White | 180 | 191 | 371
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 218 | 219 | 437

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Rate
Description: The primary objective was to determine whether the combination of sublingual buprenorphine/naloxone (SL BUP/NAL) and OXD01 was superior to SL BUP/NAL alone to reduce opioid use, measured by the treatment success rate. Treatment success was defined as the subject having >/=80% of urine drug tests negative for opioids plus >/=80% of self-reports negative for illicit opioid use from Week 6 to Week 25. Each subject was evaluated as a success or failure for this metric. The percentage of subjects in each group demonstrating treatment success was tested using the Chi-square test.
  If the subject withdrew from the study, the urine drug tests and self-reports for illicit opioid use for all visits after withdrawal were imputed as positive. If the subject completed the study with missing visits, the missing urine drug tests and self-reports for illicit opioids were imputed as positive.
Time Frame: Week 6 to Week 25
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
Participants | 70 | 67
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Superiority; p = 0.7326, Chi-squared

2. Secondary Outcome: Cumulative Response Rate
Description: The cumulative response rate was calculated from Week 6 to Week 25 of treatment. Response was defined as the presence of both a negative urine drug test for opioids and a negative self-report for illicit use of opioids at a study visit. The cumulative response rate from Week 6 to Week 25 is calculated by dividing the number of responses from Week 6 to Week 25 by the total number of visits (20), and then multiplying by 100%. The outcome is expressed as the mean percent response in each treatment group. The Kolmogorov-Smirnov method was used to compare the treatment groups.
Time Frame: Week 6 to Week 25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: percent of visits with a response
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
percent of visits with a response | 41.9 (40.83) | 42.2 (38.61)
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Superiority; p = 0.7396, Kolmogorov-Smirnoff

3. Secondary Outcome: Cumulative Response Rate - Drug Test for Illicit Use of Opioids
Description: The cumulative response rate for the illicit use of opioids was calculated from Week 6 to Week 25 of treatment. Response was defined as the presence of a negative urine drug test for opioids at a study visit. The cumulative response rate from Week 6 to Week 25 is calculated by dividing the number of responses from Week 6 to Week 25 by the total number of visits (20), and then multiplying by 100%. The outcome is expressed as the mean percent response in each treatment group. The Kolmogorov-Smirnov method was used to compare the treatment groups.
Time Frame: Week 6 to Week 25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: percent of visits with a response
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
percent of visits with a response | 43.6 (41.50) | 45.0 (39.82)
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Superiority; p = 0.8710, Kolmogorov-Smirnoff

4. Secondary Outcome: Cumulative Response Rate - Self-reports of Illicit Use of Opioids
Description: The cumulative response rate was calculated from Week 6 to Week 25 of treatment. Response was defined as the presence of a negative self-report for illicit use of opioids at a study visit. The cumulative response rate from Week 6 to Week 25 is calculated by dividing the number of responses from Week 6 to Week 25 by the total number of visits (20) and then multiplying by 100%. The outcome is expressed as the mean percent response in each treatment group. The Kolmogorov-Smirnov method was used to compare the treatment groups.
Time Frame: Week 6 to Week 25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: percent of visits with a response
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
percent of visits with a response | 51.9 (41.25) | 51.3 (39.40)
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Superiority; p = 0.8816, Kolmogorov-Smirnoff

5. Secondary Outcome: Percentage of Subjects Abstinent
Description: Abstinence is defined as a subject having urine drug tests negative for opioids as well as self-reports negative for illicit use of opioids at Week 25. Positive urine drug tests or positive timeline followback (TLFB) qualified as not abstinent. Each subject was scored as abstinent or non-abstinent and the groups were compared using a chi-squared test.
Time Frame: Week 25
Population: Full analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
Participants
  Abstinent at Week 25 | 84 | 78
  Not abstinent at Week 25 | 134 | 141
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Superiority; p = 0.5281, Chi-squared

6. Secondary Outcome: Proportion of Subjects Completing the Study
Description: A study completer was defined as a subject who completed either the urine drug screen (UDS) or the self-report assessment at the Week 25 visit. The endpoint completion rate differs from the disposition completion rate because the disposition rate used the study completion definition instead of the UDS or self-report assessment at the Week 25 visit.
Time Frame: Week 25
Population: Full analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
Participants | 137 | 127
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Superiority; p = 0.2996, Chi-squared

7. Secondary Outcome: Global Clinical Impression - Severity
Description: Clinical global Impression - severity - The severity of opioid dependence was assessed at Week 13 and Week 25 using the following assessment scale:
  Considering your total clinical experience with this particular population, how mentally ill is the subject at this time?
  0 = Not assessed
  1. = Normal, not at all ill
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill subjects
Time Frame: Week 13 and Week 25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
score on a scale
  Week 13 | 2.3 (1.18) | 2.3 (1.21)
  Week 25 | 2.2 (1.15) | 2.2 (1.23)

8. Secondary Outcome: Clinical Global Impression - Improvement
Description: Clinical global impression - improvement - Improvement in severity of opioid dependence from baseline (study Day 1) was assessed by the Investigator at the visit on Week 13 and Week 25 using the following assessment scale:
  Rate total improvement whether or not, in your judgement, it is due entirely to drug treatment. Compared to his or her condition at admission to the project, how much has the subject changed?
  0 = Not assessed
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
Time Frame: Week 13 and Week 25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
score on a scale
  Week 13 | 2.5 (1.02) | 2.5 (0.99)
  Week 25 | 2.0 (1.07) | 2.2 (1.19)

9. Secondary Outcome: Opioid Cravings - Change From Baseline
Description: Cravings for opioids were assessed by the subject through the use of a visual analog scale (VAS), where 0 mm represents "no cravings" and 100 mm represents "the most intensive craving I have ever had". The baseline craving VAS assessment was collected on study Day 1 and subsequent assessments were collected at the visit on Weeks 5, 9, 13, 17, 21, and 25.
Time Frame: Day 1 (baseline) and Weeks 5, 9, 13, 17, 21 and 25.
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
score on a scale
  Day 1 (baseline) | 34.1 (29.44) | 32.4 (29.83)
  Week 5 | -7.6 (23.80) | -6.2 (25.26)
  Week 9 | -3.8 (30.02) | -7.2 (26.87)
  Week 13 | -9.0 (26.58) | -9.6 (28.32)
  Week 17 | -6.3 (25.89) | -9.2 (28.46)
  Week 21 | -9.0 (25.90) | -11.8 (29.49)
  Week 25 | -12.0 (26.95) | -16.6 (32.13)

10. Secondary Outcome: Cumulative Response Rate - Illicit Non-opioid Drugs of Abuse
Description: The cumulative response rate was calculated from Week 6 to Week 25 of treatment. Response was defined as the presence of both a negative urine drug test for opioids and a negative self-report for illicit use of non-opioid drugs of abuse at a study visit. The cumulative response rate from Week 6 to Week 25 is calculated by dividing the number of responses from Week 6 to Week 25 by the total number of visits (20) and then multiplying by 100%. The outcome is expressed as the mean percent response in each treatment group. The Kolmogorov-Smirnov method was used to compare the treatment groups.
Time Frame: Week 6 to Week 25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: percent of visits with a response
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
percent of visits with a response | 39.31 (39.879) | 40.82 (37.625)
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Superiority; p = 0.7201, Kolmogorov-Smirnoff

11. Secondary Outcome: Resource Use - Number of Hospitalizations
Description: Number of subject hospitalizations weeks 1-25.
Time Frame: Weeks 1-25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
hospitalizations | 0.0 (0.19) | 0.0 (0.22)

12. Secondary Outcome: Resume Productive Activity
Description: Subjects were asked if they were able to resume work, school, or other productive activities. The possible responses were Yes, No, and No Change. Only subjects with non-missing data in each group were included in the analysis.
Time Frame: Week 25
Population: Full analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 179 | 165
Participants
  Yes | 97 | 107
  No | 6 | 4
  No change | 76 | 54
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Summary statistics are presented; Test type: Other; Summary statistics are presented

13. Secondary Outcome: Resource Use - Emergency Department Visits
Description: Number of subject emergency department visits weeks 1-25.
Time Frame: Weeks 1-25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: number of emergency department visits
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
number of emergency department visits | 0.1 (0.49) | 0.2 (0.55)

14. Secondary Outcome: Overdose Events
Description: Overdose events
Time Frame: Weeks 1-25
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: overdose events
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
Number analyzed (Participants) | 218 | 219
overdose events | 0.0 (0.23) | 0.0 (0.13)
Statistical Analysis 1: Comparison: SL BUP/NAL SOC Background Therapy vs SL BUP/NAL SOC Background Therapy + OXD01; Test type: Other; Summary statistics are presented

ADVERSE EVENTS:
Time Frame: 25 weeks
Arm/Group | SL BUP/NAL SOC Background Therapy | SL BUP/NAL SOC Background Therapy + OXD01
All-Cause Mortality (participants affected / at risk) | 1/218 | 0/219
Serious Adverse Events (participants affected / at risk) | 9/218 | 7/219
Other Adverse Events (participants affected / at risk) | 41/218 | 38/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SL BUP/NAL SOC Background Therapy (N=218) | SL BUP/NAL SOC Background Therapy + OXD01 (N=219)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SL BUP/NAL SOC Background Therapy (N=218) | SL BUP/NAL SOC Background Therapy + OXD01 (N=219)
COVID-19 (Infections and infestations) | 10 (10) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (4)
Nausea (Gastrointestinal disorders) | 6 (6) | 7 (7)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Anxiety (Psychiatric disorders) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 5 (6)

LIMITATIONS AND CAVEATS:
The frequent number of site visits, interactions with the Investigators and site staff, and the general level of caregiving was elevated in comparison to the routine care provided outside of a randomized and controlled clinical trial. The design of this study may not have been optimal for testing this digital therapeutic in this population and may be considered a limitation to be avoided in future clinical studies of OXD01.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04948307/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04948307/SAP_001.pdf